CLINICAL TRIAL: NCT05943665
Title: An Open Label, Phase 2, Single-arm Pilot Study to Investigate the Safety and Preliminary Effectiveness of MDMA-assisted Therapy in Veterans With Co-occurring Alcohol Use Disorder and Post-traumatic Stress Disorder (AUD-PTSD)
Brief Title: MDMA for AUD/PTSD Comorbidity
Acronym: MDMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Carolina L Haass-Koffler (Other)
Responsible Party: Sponsor-Investigator, Carolina L Haass-Koffler, Associate Professor, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000023
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder; Post Traumatic Stress Disorder
Keywords: AUD; PTSD
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MDMA-AT (Experimental): Participant will receive MDMA administration with assisted therapy (AT) by trained clinicians
  Interventions: Drug: MDMA

INTERVENTIONS:
Drug: MDMA — medication and therapy combined
  Other Names: Assisted Therapy (AT)

SUMMARY:
The study investigators are conducting the first open label pilot trial of MDMA-assisted therapy (MDMA-AT) with a comorbid sample of military veterans with a comorbid diagnosis of Alcohol Use Disorder (AUD) and Post-Traumatic Stress Disorder (PTSD). This novel experimental treatment package consists of two once-monthly Experimental Sessions of therapy combined with a divided-dose of MDMA HCl, along with non-drug preparatory and integrative therapy. The Primary Outcome measure, the Timeline Follow-back (TLFB), will evaluate changes in alcohol use over time. Changes in PTSD symptoms will also be evaluated.

DETAILED DESCRIPTION:
The study will use a longitudinal design to conduct an open label pilot trial of MDMA-AT. The study will also collect neuroimaging and biomarker data to examine brain changes pre-post treatment. Eligible participants will complete an in-person baseline assessment, undergo optional imaging protocols (if participant agrees and is medically safe to do so), engage in MDMA-AT with clinicians trained by MAPS PBC, and complete assessments at the post-treatment follow-up For complete description of the investigational plan, please the attached Clinical Protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Are able to provide proof of veteran status.
2. Are fluent in speaking and reading English.
3. At Baseline, meet criteria for Alcohol Use Disorder as measured by the SCID-5.
4. Able to safely abstain from alcohol for at least 48 hours without requiring medical detox.
5. At Baseline meet DSM-5 criteria for current PTSD with a symptom duration of at least 6 months.
6. At Baseline, have a PCL-5 score of 33 or greater.
7. At Baseline, have a confirmed PTSD diagnosis per the CAPS-5 and a Total Severity Score of 28 or greater.
8. Are able to swallow pills.
9. Agree to have study visits recorded, including Experimental Sessions, assessments, and non-drug therapy sessions.
10. Able to provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming unwell or unreachable.
11. Able to identify appropriate support person(s) to stay with the participant on the evenings of the Experimental Sessions, see Section Support Person.

    Weight
12. Body weight of at least 45 kilograms (kg). Participants with a body weight of 45 to 48 kg must also have a body mass index (BMI) within the range of 18 to 30 kg/m2.

    Sex and Contraceptive/ Barrier Requirements
13. For participants assigned female sex at birth:

    * A participant is eligible to participate if not pregnant, not planning to become pregnant, or is not breastfeeding and one of the following conditions applies
    * Is not able to become pregnant
    * Is a person able to be pregnant (PABP) and using a contraceptive method that is highly effective, with a failure rate of <1%. The investigator will evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first does of study intervention. A PABP must have a highly sensitive negative urine pregnancy test at study entry and prior to each Experimental Session, see Schedule of Activities. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a participant with an early undetected pregnancy.

    Informed Consent
14. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

    Other Inclusions
15. Agree to inform the investigators within 48 hours of any medical conditions and procedures.
16. May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
17. Participants must have a plan, agreed upon by investigator, therapy team, and study clinician, to reduce use of substances and to manage symptoms without self-medicating. Enrollment will require that, in the judgment of the investigator, therapy team, and study physician, the plan for decreasing substance use is realistic and has a good chance of succeeding to prevent substance use from impacting the safety or efficacy of the investigational treatment.
18. May have a history of or current Diabetes Mellitus (Type 2) if additional screening measures rule out underlying cardiovascular disease, if the condition is judged to be stable on effective management, and with approval by the study clinician.
19. May have hypothyroidism if taking adequate and stable thyroid replacement medication.
20. May have a history of, or current, glaucoma if approval for study participation is received from an ophthalmologist.

Exclusion Criteria:

Medical Conditions

1. Have symptomatic liver disease or have significant liver enzyme elevations.

   * Alanine transaminase (ALT) or aspartate transaminase (AST) > 3 x upper limit of normal (ULN).
   * Total bilirubin > 1.5 x ULN or direct bilirubin < 35%.
2. Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.

   • Note: Stable chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B (e.g., the presence of hepatitis B surface antigen or positive hepatitis C antibody test result without evidence of active infection at screening or within 3 months prior to starting study intervention) is acceptable if the participant otherwise meets entry criteria.
3. Have a history of seizures or delirium tremens (DTs).
4. Significant alcohol withdrawal symptoms, defined as a Clinical Institute Withdrawal Assessment of alcohol scale, revised (CIWA-Ar) >10.
5. Have a recent history of clinically significant hyponatremia or hyperthermia.
6. Have a marked Baseline QTcF interval >450 ms demonstrated on repeated ECG assessments. Participants whose QTcF exceeds this value during screening may be initially enrolled if a pre-study concomitant medication is suspected to be prolonging the QT-interval. ECGs should be repeated after initial enrollment and tapering off the pre-study concomitant medication to ensure the participant meets eligibility criteria prior to enrollment confirmation and to IMP dosing.

   • Note: The QTcF is the QT interval corrected for heart rate according to Fridericia's formula. It is either machine-read or manually over-read.
7. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate. This includes, but is not limited to, a history of myocardial infarction, cerebrovascular accident, heart failure, severe coronary artery disease, or aneurysm.

   * Participants with other mild, stable chronic medical problems may be enrolled if the study clinician and principal investigators agree the condition would not significantly increase the risk of MDMA administration or be likely to produce significant symptoms during the study that could interfere with study participation or be confused with side effects of the IMP.
   * Examples of stable medical conditions that could be allowed include, but are not limited to, Diabetes Mellitus (Type 2), Human Immunodeficiency Virus (HIV) infection, Gastroesophageal Reflux Disease (GERD), hypothyroidism (if taking adequate and stable thyroid replacement medication), glaucoma (if approval for study participation is received from an ophthalmologist). Any medical disorder judged by the investigator to significantly increase the risk of MDMA administration by any mechanism would require exclusion.
8. Have a diagnosis of controlled or uncontrolled hypertension, defined as repeated blood pressure readings of ≥ 140 millimeters of Mercury [mmHg] systolic or ≥ 90 mmHg diastolic. The diagnosis may be confirmed by repeated clinic measurements or home blood pressure monitoring if clinically indicated.
9. Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
10. Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
11. Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening.

    • Participants with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia or any other arrhythmia associated with a bypass tract may be enrolled only if they have been successfully treated with ablation and have not had recurrent arrhythmia for at least one year off all antiarrhythmic drugs or are under adequate and stable pharmacologic treatment for atrial fibrillation for at least a year, as confirmed by a cardiologist.
12. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
13. Exclusion criteria specific to MRI: non-removable ferromagnetic materials; claustrophobia; history of head trauma or injury.

    Psychiatric Conditions
14. Have engaged in a new form of psychiatric or mental health care within 12 weeks of enrollment, including Electroconvulsive Therapy (ECT) and ketamine-assisted therapy.
15. Are currently prescribed antidepressant medications (e.g., selective serotonin reuptake inhibitors) requiring a medication taper.
16. Are currently prescribed antipsychotic medications.
17. Are likely, in the investigator's opinion and via observation during the Preparatory Period, to be re-exposed to their index trauma or other significant trauma or other significant trauma during the study.
18. Have a current moderate (not in early remission in the 3 months prior to enrollment and meets at least 5 of 11 diagnostic criteria per DSM-5) or severe cannabis use disorder within the 12 months prior to enrollment (meets at least 6 of 11 diagnostic criteria per DSM-5).

    • May have current mild cannabis use disorder (meets 3 of 11 diagnostic criteria per DSM-5) or moderate cannabis use disorder in early remission for the 3 months prior to enrollment (meets 4 or 5 of 11 diagnostic criteria per DSM-5).
19. Have an active substance use (other than cannabis) disorder at any severity within 12 months prior to enrollment.
20. Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session
21. Any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS, and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled. Any participant presenting with the following on the Baseline C-SSRS will be excluded:

    * Suicidal ideation score of 4 or greater within the last 6 months of the assessment at a frequency of once a week or more
    * Suicidal ideation score of 5 within the last 6 months of the assessment
    * Any suicidal behavior, including suicide attempts or preparatory acts, within the last 6 months of the assessment. Participants with non-suicidal self-injurious behavior may be included if approved by the study clinician.
22. Would present a serious risk to others as established through clinical interview and contact with treating psychiatrist.

    Prior/Concomitant Therapy
23. Require ongoing concomitant therapy with a psychiatric medication with exceptions described in protocol section on Concomitant Medications (refer to Appendix E: Permitted and Prohibited Medications). Therapy with SSRIs at baseline is allowed as long as approved by a physician to taper off before initiating the study procedures.
24. Current use of pharmacotherapies (i.e., naltrexone or disulfiram) to treat alcohol use.
25. Require use of concomitant medications that could prolong the QT interval during Experimental Sessions.
26. Are currently engaged in trauma-focused psychotherapy or are currently in a treatment program for SUD (self-help programs are not an exclusion).

    Prior/Concurrent Clinical Study Experience
27. Current enrollment in any other clinical study involving an investigational study treatment or any other type of medical research, unless approved by the study clinician.

    Diagnostic Assessments
28. Have a history of or a current primary psychotic disorder, bipolar affective disorder type I or dissociative identity disorder assessed via the DDIS and clinical interview.
29. Have a current eating disorder with compensatory behaviors.
30. Have current major depressive disorder with psychotic features.
31. Have current Personality Disorders (paranoid, schizoid, schizotypal, antisocial, borderline, histrionic, narcissistic, avoidant, dependent, obsessive-compulsive) assessed via the SCID-5-PD. Diagnoses will be confirmed by clinical interview.

    Other Exclusions
32. Are not able to provide adequate informed consent.
33. Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the sponsor-investigator or study clinician, contraindicates participation in the study.
34. Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders.
35. Lack of social support or lack a stable living situation since the inclusion of a support person to assist the participant following Experimental Sessions is important for ensuring participant safety. If a participant is not able to identify a support person whom the research team may contact they will not be enrolled.
36. Previous participation in a MAPS-sponsored MDMA clinical trial.
37. Employees (and their immediate family members) of MAPS, MAPS Public Benefit Corporation, or MAPS Europe B.V; or individuals in a personal relationship with the sponsor investigator.
38. Have any current problem which, in the opinion of the sponsor-investigator or study clinician, might interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of standard unit drinks form the TLFB | From baseline to post-treatment follow up (18 weeks)
  Amount of alcohol consumed
CAPS score reduction | From baseline to post-treatment follow up (18 weeks)
  Severity score past 30 days

SECONDARY OUTCOMES:
Safety and tolerability | From baseline to post-treatment follow up (18 weeks)
  Number of Adverse Events
Safety and tolerability | From baseline to post-treatment follow up (18 weeks)
  Severity of Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Eaton E, Capone C, Gully BJ, Brown ZE, Monnig M, Worden MS, Swift RM, Haass-Koffler CL. Design and methodology of the first open-label trial of MDMA-assisted therapy for veterans with post-traumatic stress disorder and alcohol use disorder: Considerations for a randomized controlled trial. Contemp Clin Trials Commun. 2024 Jul 20;41:101333. doi: 10.1016/j.conctc.2024.101333. eCollection 2024 Oct. PMID 39262902